CLINICAL TRIAL: NCT02750267
Title: Closed-Loop Control in Young Children 5-8 Years Old Using DiAs Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Mark DeBoer, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18888
Record Dates: First submitted 2016-04-15; First posted 2016-04-25 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes Mellitus (T1DM); Artificial Pancreas Project (APP); Diabetes Assistant (DiAs); Closed-Loop Control (CLC); Continuous Glucose Monitor; Pediatric; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): In this randomized, cross-over study, the intervention involves blood glucose control using a Closed Loop system run by the Diabetes Assistant (DiAs) during a stay at a Research House/Hotel. All subjects will have blood glucose data compared between their usual diabetes care (at home, using home insulin pump) and this Closed-Loop care (at Research House/Hotel using the DiAs system). Subjects who are randomized to Group A will have home care evaluated before the Research House/Hotel admission. Subjects in this arm will participate in CGM training and data collection prior to the Research House/Hotel admission.
  Interventions: Device: Diabetes Assistant (DiAs) with Closed-Loop
- Group B (Experimental): Group B is identical to Group A with the exception that usual diabetes care (at home, using home insulin pump) will be evaluated after the Research House/Hotel admission. Subjects who are randomized to Group B will participate in CGM training and data collection after the Research House/Hotel admission. As with Group A, all subjects will use Diabetes Assistant (DiAs) with Closed-Loop during the admission.
  Interventions: Device: Diabetes Assistant (DiAs) with Closed-Loop

INTERVENTIONS:
Device: Diabetes Assistant (DiAs) with Closed-Loop — All subjects will use DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a Research House/Hotel admission that will last up to 72 hours.

SUMMARY:
The overall aim of this proposed research is to determine the safety, feasibility and efficacy (AP vs at home use of SAP) of the Diabetes Assistant (DiAs) controller in day and night closed-loop control in young children 5-8 years old with type 1 diabetes over multiple 48 hours in an out-patient setting.

DETAILED DESCRIPTION:
Young children with Type 1 Diabetes (T1D) in the age range of 5-8 years old are a population with clear needs but unique challenges regarding the application of artificial pancreas (AP) technologies. Young children are likely to benefit from an AP system, with current deficits in glycemic control that include both significant hypoglycemia and sub-optimal HbA1c levels; however, they have undeveloped abilities to control and interact with the AP system, posing potential safety issues. During the hours that these children are away from their parents at school and elsewhere, they lack the sophistication to operate the currently-available tools in an AP system--and may induce harm if they are allowed to do so, causing parental resistance to AP use. Commercially-available insulin pumps have mechanisms to lock access to children to prevent inappropriate insulin-delivery. However, the AP is more complex than an insulin pump, both in requiring more detailed setting information (that a child could adversely alter) and in providing alerts for impending low- and high-blood glucose (BG) levels (that one wouldn't want to lock out to child use). These functions are all run via a platform on a smart phone-a device with which young children may already feel a high degree of familiarity and thus be more likely to attempt to explore and potentially change settings. It is likely that young children will benefit the most from a system that gives them access to some AP features but provides access to other features only for their parents. In this sense, young children require a device that is not user-centered as much as family-centered. A redesign of the system to provide appropriate access to AP tools-in which certain users can obtain access to certain functionalities-is direly needed before children in this age range can benefit from the improvements in blood glucose (BG) control that the AP has to offer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes,

  * The diagnosis of type 1 diabetes is based on the investigator's judgment
  * C peptide levels and antibody determinations are not required
* Daily insulin therapy for ≥ 12 months
* Insulin pump therapy for ≥ 3 months
* Age ≥5 - ≤8 years old
* Avoidance of acetaminophen-containing medications (i.e. Tylenol) while wearing the continuous glucose monitor.
* Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

* Diabetic ketoacidosis in the past month
* Hypoglycemic seizure or loss of consciousness in the past 3 months
* History of seizure disorder (except for hypoglycemic seizure)
* History of any heart disease including coronary artery disease, heart failure, or arrhythmias
* Cystic fibrosis
* Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria).
* Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir or Glargine).
* Subjects requiring other anti-diabetic medications other than insulin (oral or injectable).
* Presence of a febrile illness within 24 hours of admission or acetaminophen use while wearing the CGM. The subject may be rescheduled for Research House/Hotel Admission if these criteria are not met. The study subject will not participate in the trial if these conditions are met.
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal insufficiency

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. DeBoer, MD, Principal Investigator — University of Virginia, Pediatrics, Endocrinology/Diabetes
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Not yet determined

REFERENCES:
- [Background] DeBoer MD, Breton MD, Wakeman C, Schertz EM, Emory EG, Robic JL, Kollar LL, Kovatchev BP, Chernavvsky DR. Performance of an Artificial Pancreas System for Young Children with Type 1 Diabetes. Diabetes Technol Ther. 2017 May;19(5):293-298. doi: 10.1089/dia.2016.0424. Epub 2017 Apr 20. PMID 28426239
- See also: Use of an AP in young children was safe and resulted in improved mean BG without increased hypoglycemia. This suggests that AP use in young children is safe and improves overall diabetes control. — https://www.ncbi.nlm.nih.gov/pubmed/28426239

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A- Home Care Before Closed-Loop Control: In this randomized, cross-over study, the intervention involves blood glucose control using a Closed Loop system run by the Diabetes Assistant (DiAs) during a stay at a Research House/Hotel. All subjects will have blood glucose data compared between their usual diabetes care (at home, using home insulin pump) and this Closed-Loop care (at Research House/Hotel using the DiAs system). Subjects who are randomized to Group A will have home care evaluated before the Research House/Hotel admission. Subjects in this arm will participate in CGM training and data collection prior to the Research House/Hotel admission.
  Diabetes Assistant (DiAs) with Closed-Loop: All subjects will use DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a Research House/Hotel admission that will last up to 72 hours.
- Group B- Closed-Loop Control Before Home Care: Group B is identical to Group A with the exception that usual diabetes care (at home, using home insulin pump) will be evaluated after the Research House/Hotel admission. Subjects who are randomized to Group B will participate in CGM training and data collection after the Research House/Hotel admission. As with Group A, all subjects will use Diabetes Assistant (DiAs) with Closed-Loop during the admission.
  Diabetes Assistant (DiAs) with Closed-Loop: All subjects will use DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a Research House/Hotel admission that will last up to 72 hours.
Period: Overall Study
Arm/Group | Group A- Home Care Before Closed-Loop Control | Group B- Closed-Loop Control Before Home Care
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A- Home Care Before Closed-Loop Control | Group B- Closed-Loop Control Before Home Care | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7 [6.25 to 7.75] | 7 [7 to 7] | 7 [6.75 to 7.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
HbA1c [Median (Inter-Quartile Range); unit: percentage of HbA1C] | 7.7 [7.2 to 7.8] | 7.6 [7.1 to 7.8] | 7.7 [7.1 to 7.8]
Diabetes Duration [Median (Inter-Quartile Range); unit: years] | 4.9 [2.2 to 6.1] | 3.3 [3.2 to 5.0] | 3.7 [2.9 to 5.7]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Sensor Glucose Readings Between 70-180 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: percentage of time in range
Groups:
- Home Care (Pump+CGM): All 12 subjects completed 68 hours of usual, home care using their home insulin pumps and a study CGM. The 6 subjects in Group A completed the home care portion before the Hotel admission, and the 6 subjects in Group B completed the home care portion after the Hotel admission.
- Diabetes Assistant (DiAs) With Closed-Loop Control: All 12 subjects used the DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a 68 hour Hotel admission.
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
percentage of time in range | 46.9 (2.7) | 73.1 (2.7)

2. Secondary Outcome: Percent of Time Sensor Glucose Readings Are <70 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: percentage of time below 70 mg/dL
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
percentage of time below 70 mg/dL | 1.6 (1.2) | 1.1 (1.1)

3. Secondary Outcome: Percent of Time Sensor Glucose Readings Are >150 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Groups:
- Home Care (Pump+CGM): All 12 subjects completed 68 hours of usual, home care using their home insulin pumps and a study CGM. The 6 subjects in Group A completed the home care portion before the Hotel admission, and the 6 subjects in Group B completed the home care portion after the Hotel admission. The current secondary outcome was not specifically analyzed.
- Diabetes Assistant (DiAs) With Closed-Loop Control: All 12 subjects used the DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a 68 hour Hotel admission. The current secondary outcome was not specifically analyzed.
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percent of Time Sensor Glucose Readings Are >180 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: percentage of time above 180 mg/dL
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
percentage of time above 180 mg/dL | 51.5 (0.8) | 25.8 (2.8)

5. Secondary Outcome: Percent of Time Sensor Glucose Readings Are >250 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: percentage of time above 250 mg/dL
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
percentage of time above 250 mg/dL | 20.8 (9.9) | 6.3 (5.4)

6. Secondary Outcome: Percent of Time Sensor Glucose Readings Are >400 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Distribution of Sensor and Meter Glucose Values (Maximum, Minimum, Median, Interquartile Range, Mean, Standard Deviation)
Description: All subjects have CGM and handheld glucose meter output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Distribution of Sensor and Meter Glucose Values (Maximum)
Description: as for outcome 7
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Distribution of Sensor and Meter Glucose Values (Minimum)
Description: as for outcome 7
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Distribution of Sensor and Meter Glucose Values (Median/Interquartile Range)
Description: as for outcome 7
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Mean BG (as Measured by CGM)
Description: as for outcome 7
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
mg/dL | 190 (7.4) | 152 (4.2)

12. Secondary Outcome: Hypoglycemia Area Under the Curve <60
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Hypoglycemia Area Under the Curve <70 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Hyperglycemia Area Under the Curve >180
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Hyperglycemia Area Under the Curve >250 mg/dL
Description: All subjects have CGM output analyzed and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Incidence of Hypoglycemia Per Subject, Defined by Handheld Meter Glucose <70 mg/dL
Description: All subjects have hypoglycemia monitored by meter analysis and compared between time on closed-loop system and time on usual care period.
Time Frame: 68 hours
Measure: Mean (Standard Deviation); unit: events per subject, glucometer <70mg/dL
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 12 | 12
events per subject, glucometer <70mg/dL | 4.0 (1.0) | 3.3 (1.0)

17. Secondary Outcome: End of Night Blood Glucose
Description: All subjects have blood glucose evaluated upon rising (approximately 7 am) and compared between time on closed-loop system and time on usual care period.
Time Frame: 72 hours
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collect over two 72 hour periods for each subject. Over the entire study, adverse events were collected over a 216 hour period (Group A's 72 hr home period, 72 hr hotel period, Group B's 72 hr home period).
Groups:
- Diabetes Assistant (DiAs) With Closed-Loop Control: All 12 subjects used the DiAs Medical Platform, a study insulin pump and continuous glucose monitor (CGM) in closed-loop mode during a 68 hour Hotel admission. The 6 subjects in Group A completed the home care portion before the Hotel admission, and the 6 subjects in Group B completed the home care portion after the Hotel admission.
Arm/Group | Home Care (Pump+CGM) | Diabetes Assistant (DiAs) With Closed-Loop Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Care (Pump+CGM) (N=12) | Diabetes Assistant (DiAs) With Closed-Loop Control (N=12)
Sore Knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes